CLINICAL TRIAL: NCT03392792
Title: Regisry of the Stroke Patients in Assiut University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noura Abdel hakim abdel Mohsen, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Assiut u
Record Dates: First submitted 2017-12-14; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: All Patients With Ischemic Cerebrovascular Stroke Aged ≥18 Years of Both Sex
MeSH Terms: interventions — Tissue Plasminogen Activator; Thrombectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tissue plasmnogen activator (Active Comparator)
  Interventions: Drug: tissue plasminogen activator
- thrombectoy (Active Comparator)
  Interventions: Procedure: thrombectomy

INTERVENTIONS:
Drug: tissue plasminogen activator — role of tissue plasminogen activator in patient with acute ischemic stroke having selective criteria for rTPA
  Other Names: rtpa
  Arms: tissue plasmnogen activator
Procedure: thrombectomy — role of thrombectomy in patient with acute ischemic stroke
  Arms: thrombectoy

SUMMARY:
• Aim of the work To register all type of acute stroke admitted in Assiut university Hospital and assessment of their risk factor, morbidity and Mortality

ELIGIBILITY:
Inclusion Criteria:

* All patients with stroke aged ≥18 years of both sex
* Written consent was taken for all patient either from the patient himself of closes relative after explaning to them the type of treatment benefits and possible risks

Exclusion Criteria:

* Stroke due to metabolic causes as hypoglycemia liver, Renal failure and other metabolic causes
* Stroke due to Brain tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Registry of the stroke Patients in Assist University Hospital | one year